CLINICAL TRIAL: NCT00004126
Title: A Phase II Study of Oxaliplatin in Combination With Paclitaxel in Non-Small Cell Lung Cancer
Brief Title: Paclitaxel and Oxaliplatin in Treating Patients With Recurrent or Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10014; UCCRC-10014; NCI-T99-0008
Record Dates: First submitted 1999-12-10; First posted 2004-05-21 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Oxaliplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental): Paclitaxel 175 mg/m2 : administered by 1-hour constant rate IV infusion through a pump on day 1 of each cycle. Oxaliplatin 130 mg/m2 : On Day 1 of each 21-day treatment cycle, patients receive oxaliplatin diluted in 250-500 mL Dextrose 5% in Water infused intravenously over 2 hours.
  Interventions: Drug: oxaliplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: oxaliplatin
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining paclitaxel and oxaliplatin in treating patients who have recurrent or advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the overall, partial, and complete response rates in patients with advanced non-small cell lung cancer treated with oxaliplatin plus paclitaxel. II. Assess the overall survival, time to tumor progression, and toxicities associated with this combination regimen in this patient population. III. Assess the neurologic toxicity of this combination regimen and its correlation with creatinine clearance in these patients.

OUTLINE: This is a multicenter study. Patients receive paclitaxel IV over 1 hour followed by oxaliplatin IV over 2 hours on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients are followed for at least 2 years or until death.

PROJECTED ACCRUAL: Approximately 17-37 patients will be accrued for this study within 24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed non-small cell lung cancer (NSCLC) Stage IIIB with pleural effusion OR Stage IV OR Recurrent disease Bidimensionally measurable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Karnofsky 50-100% Life expectancy: Not specified Hematopoietic: WBC greater than 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin normal SGOT less than 2 times normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 50 mL/min BUN less than 1.5 times normal Cardiovascular: No symptomatic congestive heart failure No unstable angina or myocardial infarction within the past 6 months No evidence of heart block greater than first degree, bundle branch block, or ventricular or supraventricular arrhythmia Other: No allergy to platinum compounds or antiemetics appropriate for study No other uncontrolled illness No active or ongoing infection No evidence of peripheral neuropathy by physical exam or history Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 6 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for advanced NSCLC At least 4 weeks since prior chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: Not specified Other: No other concurrent investigational agents No concurrent antiretroviral therapy for HIV positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 1999-11; Primary Completion 2001-01 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Ann M. Mauer, MD, Study Chair — University of Chicago
Locations (11):
- United States (11):
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Cancer Care Specialists of Central Illinois, S.C., Decatur, Illinois
  - Evanston Northwestern Health Care, Evanston, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Michiana Hematology/Oncology P.C., South Bend, Indiana
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio

REFERENCES:
- [Result] Winegarden JD, Mauer AM, Otterson GA, Rudin CM, Villalona-Calero MA, Lanzotti VJ, Szeto L, Kasza K, Hoffman PC, Vokes EE; University of Chicago Phase II Network; Ohio State University. A phase II study of oxaliplatin and paclitaxel in patients with advanced non-small-cell lung cancer. Ann Oncol. 2004 Jun;15(6):915-20. doi: 10.1093/annonc/mdh215. PMID 15151948